CLINICAL TRIAL: NCT04204655
Title: Investigation of the Influence of the Body Composition of Neurological (Early) Rehabilitants as Well as Their Change in the Course of Rehabilitation and the Effect on Rehabilitation Success - a Pilot Study
Brief Title: Influence of the Body Composition of Neurological (Early) Rehabilitants on Rehabilitation Success
Status: Active, not recruiting | Type: Observational
Sponsor: BDH-Klinik Hessisch Oldendorf (Other)
Responsible Party: Sponsor
Other Study IDs: BIA-Studie
Record Dates: First submitted 2019-12-13; First posted 2019-12-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Neurological Rehabilitation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Cohort: rehabilitants of the phase B, C and D during neurological rehabilitation
  Interventions: Diagnostic Test: BIA

INTERVENTIONS:
Diagnostic Test: BIA — Bioelectrical Impedance Analysis

SUMMARY:
An optimal nutritional supply is associated with better outcome and recovery. For investigating the influence of the nutritional status and body composition on the course of rehabilitation, bioelectrical impedance analyzes (BIA) should be carried out on neurological (early) rehabilitants during the rehabilitation process.

Possible disturbances, suitable outcome valuesfor evaluation of the rehabilitation success (depending on the rehabilitation phase) as well as the required frequency of the BIA measurements in rehabilitation should be estimated with the help of this pilot study.

DETAILED DESCRIPTION:
An optimal coverage of the required calorie requirement is a basic prerequisite for a speedy recovery. One study reports that almost every fourth patient is malnourished in German hospitals. Malnutrition is in turn associated with more complications, higher mortality and longer length of stay. The current DGEM (Deutsche Gesellschaft für Ernährungsmedizin) guideline "Clinical nutrition in intensive care" recommends a calorie intake of 24 kcal per kg body weight during the acute phase of the disease (days 1 to 7) and an increase of calorie intake to 36 kcal per kg body weight in the convalescence and rehabilitation phase.

In a recent study evaluating the weight profile of neurological, enteric-coated early rehabilitants in rehabilitation, 60.6% of patients had weight loss during rehabilitation. Men were also more likely to lose weight than women. In addition, the caloric care of "underweight patients" had a decisive influence on the neurological outcome (as measured by the early rehab barthel-index(FRBI)). For example, underweight patients who were under-served showed significantly lower improvements in FRBI than underweight patients who were over-served.

In another study, the weight of patients remained stable through the use of a nutritional assessment tool (EAT). Also the gender difference was not confirmed in the group with the EAT. The weight change in the rehabilitation course correlated significantly with the difference between the calculated and the average calories received per day. However, an effect of EAT on the frequency of complications or the neurological outcome could not be demonstrated in this study.

However, as body weight may be affected by water balance (edema) and gastrointestinal complications such as constipation, vomiting and diarrhea, consideration of body weight to check diet / nutrition status alone is insufficient. Qualitative statements such as an increase / decrease in muscle mass can not be made on the basis of the weight data. Therefore, in the planned pilot study body composition will be documented by means of bioelectric impedance analysis (BIA) in neurological (early) rehabilitants during rehabilitation. At the same time, various outcome parameters are to be recorded.

The aim of this pilot study is to identify the number and frequency of BIA measurements required to assess the status of care. On the basis of this data, a study is then to be designed to investigate the success of rehabilitation as a function of nutritional status and muscle mass.

ELIGIBILITY:
Inclusion Criteria:

* neurological disease

Exclusion Criteria:

* electrical implant as cardiac pacemaker, medications pumps, defibrillators
* pregnancy or breastfeeding period
* take part on another study within the last 30 days
* spasticity
* amputation of limbs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Included in each case are 15 neurological and neurosurgical (early) rehabilitants of phase B, C and D (45 patients in total) of both sexes aged ≥ 18 years.
Sampling Method: Non-Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2019-11-25 (Actual); Primary Completion 2023-09-25 (Actual); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Functional Status | 3 minutes
  The Early Rehabilitation Barthel Index were determined upon admission and at the end of rehabilitation.
Disabilities | 3 minutes
  An ICF-Assessment of 20 items is used for determination of disabilities of activities and body functions. The severity of each item is scored from zero ("no impairment") to four ("complete impairment") upon admission and at the end of rehabilitation.
Muscle Strenght | 3 minutes
  The hand force is measured with a hand force dyometer three times on each hand upon admission and at the end of rehabilitation.
Mobility | 4 minutes
  The mobility is assed by the Rivermead Mobility Index.
Lenght Of Stay | < 1 minute
  duration of neurological rehabilitation (in days)
Mortality | < 1 minute
  Number of deaths
Discharge Level | < 1 minute
  Status at discharge (discharged at home / long-term care facility, follow-up rehabilitation, death, transfer to acute hospital)

SECONDARY OUTCOMES:
Bioelectrical Impedance | 15 minutes
  Bioelectrical Impedances for all body segments: right arm, left arm, right leg, left leg, trunk, right body side and left body side.
Nutritional Risk Screening (NRS 2002) | 5 minutes
  Malnutrition upon admission and at discharge is assed by the Nutritional Risk Screening (NRS 2002).
Mini Nutritional Assessment (MNA) | 5 minutes
  Malnutrition upon admission and at discharge is assed by the Mini Nutritional Assessment (MNA).

OTHER OUTCOMES:
Blood Pressure | 1 minute
  Blood pressure (mmHg) is measured before each BIA measurement.
Pulse | < 1 minute
  Pulse (bmp) is measured with a finger pulse oxymeter before each BIA measurement.
Saturation | < 1 minute
  Saturation (%) is measured with a finger pulse oxymeter before each BIA measurement.
Body Height | 2 minutes
  Height is measured in a standing position with a measuring tape. In the case that the patient is not able to stand, the measurement is performed in a lying position.
Body weight | 5 minutes
  Weight (kg) is measured in the morning with clothes but without shoes.
Hip Circumference | 1 minute
  Hip circumference is measured with a measuring tape in a standing position (or lying position if the patient can not stand).
Waist Circumference | 1 minute
  Waist circumference is measured with a measuring tape in a standing position (or lying position if the patient can not stand).
Calf Circumference | 1 minute
  Calf circumference is measured with a measuring tape in a standing position (or lying position if the patient can not stand).

CONTACTS AND LOCATIONS:
Overall Officials: Jens D Rollnik, Prof. Dr., Study Director — BDH-Klinik Hessisch Oldendorf
Locations (1):
- Institute for Neurorehabilitation Research, BDH-Clinic Hessich Oldendorf, Hessisch Oldendorf, Lower Saxony, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pirlich M, Schutz T, Norman K, Gastell S, Lubke HJ, Bischoff SC, Bolder U, Frieling T, Guldenzoph H, Hahn K, Jauch KW, Schindler K, Stein J, Volkert D, Weimann A, Werner H, Wolf C, Zurcher G, Bauer P, Lochs H. The German hospital malnutrition study. Clin Nutr. 2006 Aug;25(4):563-72. doi: 10.1016/j.clnu.2006.03.005. Epub 2006 May 15. PMID 16698132
- [Background] Sorensen J, Kondrup J, Prokopowicz J, Schiesser M, Krahenbuhl L, Meier R, Liberda M; EuroOOPS study group. EuroOOPS: an international, multicentre study to implement nutritional risk screening and evaluate clinical outcome. Clin Nutr. 2008 Jun;27(3):340-9. doi: 10.1016/j.clnu.2008.03.012. Epub 2008 May 27. PMID 18504063
- [Background] Elke G, Hartl WH, Kreymann KG, Adolph M, Felbinger TW, Graf T, de Heer G, Heller AR, Kampa U, Mayer K, Muhl E, Niemann B, Rumelin A, Steiner S, Stoppe C, Weimann A, Bischoff SC. [DGEM Guideline "Clinical Nutrition in Critical Care Medicine" - short version]. Anasthesiol Intensivmed Notfallmed Schmerzther. 2019 Jan;54(1):63-73. doi: 10.1055/a-0805-4118. Epub 2019 Jan 8. German. PMID 30620956
- [Background] Schmidt SB, Boltzmann M, Rollnik JD. Nutritional situation of enterally fed patients in neurological early rehabilitation and impact of nutritional status on functional outcome. Clin Nutr. 2020 Feb;39(2):425-432. doi: 10.1016/j.clnu.2019.02.011. Epub 2019 Feb 10. PMID 30799195
- [Background] Schmidt SB, Boltzmann M, Krauss JK, Stangel M, Gutenbrunner C, Rollnik JD. Standardized nutritional supply versus individual nutritional assessment: Impact on weight changes, complications and functional outcome from neurological early rehabilitation. Clin Nutr. 2020 Apr;39(4):1225-1233. doi: 10.1016/j.clnu.2019.05.013. Epub 2019 May 16. PMID 31151820
- [Background] Stucki G, Cieza A, Geyh S, Battistella L, Lloyd J, Symmons D, Kostanjsek N, Schouten J. ICF Core Sets for rheumatoid arthritis. J Rehabil Med. 2004 Jul;(44 Suppl):87-93. doi: 10.1080/16501960410015470. PMID 15370754
- [Background] Geyh S, Cieza A, Schouten J, Dickson H, Frommelt P, Omar Z, Kostanjsek N, Ring H, Stucki G. ICF Core Sets for stroke. J Rehabil Med. 2004 Jul;(44 Suppl):135-41. doi: 10.1080/16501960410016776. PMID 15370761